CLINICAL TRIAL: NCT00715390
Title: Dysrhythmias During General Anesthesia in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-10-3923
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2011-03-01 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Arrhythmias, Cardiac
Keywords: Children; Cardiac Arrhythmia; General Anesthesia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1-Children receiving anesthesia: The sample of patients screened will be the entire electronic anesthesia record database from 1998 until 2004 looking for subjects that have dysrhythmias.

SUMMARY:
To describe the types and incidence of cardiac dysrhythmias that occur under anesthesia in the present anesthesia environment.

DETAILED DESCRIPTION:
It is unclear what the current state of anesthesia associated dysrhythmias is in the pediatric population. This was last investigated retrospectively in 1992 when the predominant volatile agent used for inhalation induction was halothane. Sevoflurane was approved by the Food and Drug Administration in 1995. Since that time, Sevoflurane has displaced halothane as the agent of choice for inhalation induction and has relegated halothane to be used in a narrow niche which primarily involves patients with very specific congenital heart diseases. It has been described that halothane has a larger proarrhythmic effect than sevoflurane for ventricular dysrhythmias. With the transition from the halothane to the sevoflurane era, a reassessment of the incidence and types of dysrhythmias occurring in non-cardiac pediatric patients is important.

ELIGIBILITY:
Inclusion Criteria:

Children, while under anesthesia, having

1. circumstances of tachycardia and bradycardia,
2. administration of medications used in the treatment of dysrhythmias,
3. the commentary which includes comment about the heart rhythm or therapy for dysrhythmia,
4. in the quality assurance database for evidence of dysrhythmia

Exclusion Criteria:

Children with a known pre-operative:

1. prior history of dysrhythmia and/or
2. residual congenital heart disease
3. anti/pro dysrhythmic medications

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have undergone anesthesia at the Children's Hospital of Philadelphia or at one of CHOP's satellite surgicenters, and whose anesthetic record was recorded electronically into the Compurecord system will be screened.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald S Litman, DO, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We performed a retrospective chart review of anesthetics administered at The Children's Hospital of Philadelphia from July 1998 through July 2004.
Pre-assignment Details: Excluded were patients with known arrhythmias or pro-arrhythmic conditions, patients with congenital heart disease and patients undergoing cardiac surgery or cardiac catheterization.
Groups:
- Children With Dysrhythmia Events During Anesthesia: The sample of patients screened will be the entire electronic anesthesia record database from 1998 until 2004 looking for subjects that have dysrhythmias.
Period: Overall Study
Arm/Group | Children With Dysrhythmia Events During Anesthesia
Started | 234 (114,209 Anesthetic records were screened to identify 234 records.)
Eligible | 234
Completed | 234 (These were broken down to different types of dysrhythymia.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Children With Dysrhythmia Events During Anesthesia
Number analyzed (Participants) | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 234
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 134
Region of Enrollment [Number; unit: participants]
  United States | 234
Children with potential intraoperative dysrhythmias [Number; unit: participants] — Subjects were identified by flagging charts that included the administration of anti-arrhythmic drugs, significant variation in heart rate or pulse rate, and identification of certain keywords known to be associated with the development of an arrhythmia.
  participants | 234

OUTCOME MEASURES:

1. Primary Outcome: Arrhythmias During General Anesthesia in Children
Time Frame: July 1998 through July 2004
Measure: Number; unit: participants
Arm/Group | Children With Dysrhythmia Events During Anesthesia
Number analyzed (Participants) | 220
participants | 220

ADVERSE EVENTS:
Arm/Group | Children With Dysrhythmia Events During Anesthesia
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes